CLINICAL TRIAL: NCT06865391
Title: Multıdımensıonal Effects Of Delayed Cord Clampıng and Mılkıng on Placental Processes and Maternal-Newborn Hematologıcal Parameters ın Postpartum Cord Management
Brief Title: Multıdımensıonal Effects Of Delayed Cord Clampıng and Mılkıng on Placental Processes
Acronym: DCC&MILKHEM P
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kahramanmaras Sutcu Imam University (Other)
Responsible Party: Principal Investigator, Hatice Gul OZTAS, Principal Investigator, Kahramanmaras Sutcu Imam University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: KahramanmaraşSIUI5
Record Dates: First submitted 2025-02-14; First posted 2025-03-07 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: 18 Years and Over; Newborn Health; 37 or More Completed Weeks of Gestation
Keywords: delayed cord clamping; cord milking; placenta; clinical outcome; midwifery
MeSH Terms: interventions — Umbilical Cord Clamping

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental (Experimental): Delayed cord clamping (DCC) was defined as clamping the umbilical cord 90 seconds after birth. A stopwatch was used to record the time of all interventions and was noted in the study protocol.
  Umbilical Cord Milking (UCM) is the process of grasping the umbilical cord towards the newborn before cutting the umbilical cord and pushing the blood towards the newborn 3-4 times within 20 seconds." In this group, early cord clamping (<30 seconds) was performed after birth from 25-30 cm ahead of the newborn for a total of 4 times. UCM, with one hand, the cord was pinched and held closest to the placental end, the other hand was used to milk blood towards the infant where at the umbilical endpoint the cord was held. This served as one milking motion. The cord was then released at the placental end and allowed to refill over 1 to 2 seconds between each milking motion. This was repeated a total of 4 times. After milking, the cord was clamped and cut, and the neonate was handed over to
  Interventions: Behavioral: Delayed cord clamping
- control group (No Intervention): standart care grup

INTERVENTIONS:
Behavioral: Delayed cord clamping
  Arms: Experimental

SUMMARY:
This study was conducted to evaluate the effects of delayed cord clamping and milking the umbilical cord of term babies after 90 seconds during vaginal birth on the newborn and the mother and to determine whether it is a suitable alternative method for cord management after birth.

Methods: The study was conducted in the form of a randomized controlled design. The study was conducted in a hospital in eastern Turkiye between February -January 2025. The study was completed with 108 women who had vaginal delivery at term (DCC group n=36, UCM group n=36, control group n=36). Participants were assigned to groups by simple randomization. Data collection tools were used to collect demographic information, maternal hemoglobin, and hematocrit values, placental abruption time, newborn APGAR scores, umbilical cord pH levels, and day 7 hematological/biochemical parameters.

DETAILED DESCRIPTION:
Labor and the postpartum period are critical periods that can have long-term effects on both maternal and neonatal health. Evidence-based interventions implemented during this period play a significant role in maternal physiological recovery, placental abruption, neonatal health parameters, and long-term health bilical cord management (delayed cord clamping [DCC] and umbilical cord milking [UCM]) has become an important research topic in recent years regarding its effects on maternal and neonatal outcomes DCC is defined by clamping the umbilical cord after birth for a certain period of time, and it has been shown that this practice can increase neonatal hemoglobin and hematocrit levels and reduce the risk of neonatal anemia . At the same time, it has been reported that DCC is especially recommended to reduce iron deficiency anemia in low-income countries . However, there are also views that DCC may prolong the time to placental abruption and increase the risk of postpartum hemorrhage in the mother UCM is defined as the process of pushing blood in the umbilical cord to the newborn with mechanical movement. There are studies indicating that this method improves oxygen transport by increasing blood volume and reduces the risk of intraventricular hemorrhage while increasing cardiovascular stability in premature babiesHowever, there are conflicting results in the literature regarding the effects of this method on hyperbilirubinemia and hemoglobin increase The effects of these different methods in umbilical cord management on maternal hemoglobin and hematocrit levels, placental abruption time, neonatal hematological and biochemical parameters, and postpartum complications have been an important area of research . Studies have emphasized that there are important relationships between the duration of placental abruption and neonatal health indicators and that these processes should be examined in detail . It has been reported that providing additional blood volume, especially in premature babies, can improve neonatological parameters and have important effects on maternal health . Therefore, studies have emphasized that the relationships between the duration of placental abruption and the timing of separation signs and neonatal health indicators should be examined in detail .In this study, many outcomes such as placental abruption time, maternal hemoglobin and hematocrit levels, and neonatal hematological and biochemical parameters were evaluated in this context. Therefore, this study aims to provide evidence to make a significant contribution to the literature on umbilical cord management practices and to determine the place of these practices in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* being 18 years of age and older,
* having a single healthy newborn,
* having a 37-42 week pregnancy,
* having a baby in cephalic presentation, and
* having a first birth (nulliparous).

Exclusion Criteria:

* women with gestational anemia,
* having abnormal placentation (such as bleeding, hypertension),
* having a maternal hemorrhage,
* having Rh isoimmunization, and
* having a baby with a major congenital malformation

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — YES
Enrollment: 108 (Actual)
Dates: Start 2025-03-20 (Actual); Primary Completion 2025-03-28 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
APGAR | 5 minutes after birth
  APGAR scores,Developed in 1953 by Dr Virginia Apgar for the quantitative assessment of the vitality of the newborn, the scoring system is used in almost all neonatal units as an easy and rapid method to determine the condition of the child at birth. Its aim is to encourage closer observation and to provide a more precise assessment of the clinical status of infants. According to the Apgar scoring system, the newborn is assessed at 1 and 5 minutes after birth and if necessary, the scoring is repeated every 5 minutes. Apgar scoring is based on 5 objective parameters: 1. peak heart rate, 2. respiratory pattern, 3. muscle tone, 4. skin colour, 5. response to stimulation. Each parameter is given 0, 1 and 2 points. The scores given for each parameter are summed. Values between 710 points are considered healthy newborns, while 4-6 points are considered moderate depression and 0-3 points are considered severe depression.

CONTACTS AND LOCATIONS:
Locations (1):
- Kahramanmaraş Sütçü İmama Universty, Kahramanmaraş Merkez, K.maraş, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No